CLINICAL TRIAL: NCT02438462
Title: Evaluation of Performances of Soluble Fibrin Assay for Diagnosing Pulmonary Embolism
Brief Title: Soluble Fibrin for Diagnosing Pulmonary Embolism
Acronym: SOFIE
Status: Completed | Type: Observational
Sponsor: Diagnostica Stago R&D (Industry)
Collaborators: European Georges Pompidou Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SOFIE 2015-A00094-45
Record Dates: First submitted 2015-05-05; First posted 2015-05-08 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Pulmonary Embolism (PE)
Keywords: Pulmonary Embolism; Soluble Fibrin; D-Dimers; Clinical Probability Score; Imaging
MeSH Terms: conditions — Pulmonary Embolism | interventions — thrombus precursor protein, human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Frozen citrated Poor Platelets Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group with PE: The criteria for confirmation of PE are:
  * PE on spiral computed tomography (CT)
  * proximal deep vein thrombosis on ultrasound (US)
  * thromboembolic events objectively confirmed during the follow up
  Interventions: Other: Soluble Fibrin
- Group without PE: The criteria for exclusion of PE are:
  * low or moderate clinical probability and D-dimer ELISA <0.50 µg/mL or <10xage in patients older than 50 years and negative follow up
  * low and moderate clinical probability and negative CT and negative follow up
  * high clinical probability and negative CT, US and follow up.
  Interventions: Other: Soluble Fibrin

INTERVENTIONS:
Other: Soluble Fibrin — Calculating the area under the ROC curve of the Soluble Fibrin assay for the diagnosis of PE before evaluating the diagnostic performance of the assay.

SUMMARY:
The purpose of the study is to evaluate the performances of Soluble Fibrin for diagnosing Pulmonary Embolism. Secondary objective is to compare the diagnostic performances of the Soluble Fibrin Assay and the D-Dimer test.

DETAILED DESCRIPTION:
Rationale. Pulmonary embolism (PE) is a major public health problem. D-dimer (D-Di) assay is useful to exclude the PE but not specific, requiring irradiating and expensive imaging tests. Preliminary results suggest that the Soluble Fibrin (SF) assay has a sensitivity comparable to the D-Di one, but a higher specificity and thus would limit the use of imaging tests.

Main objective. To compute the area under the ROC curve of the Soluble Fibrin assay for the diagnosis of PE and to assess the other diagnostic characteristics of the SF assay.

Patients. Inclusion criteria: patients 18 years or older, referred to the Emergency or Respiratory and Intensive Care Medicine Units, for clinically suspected of PE.

Exclusion criteria: pregnancy, contraindication to iodinated contrast media, anticoagulant drug at curative doses, patients with suspected PE during hospitalization and those for which the three month-follow up is impossible.

The protocol was approved by the Ethics Committee on March 2015. The study will be conducted in compliance with French regulations after ethics approval.

Reference algorithm. PE has to be confirmed or excluded by the reference algorithm combining clinical probability, D-Dimer, imaging tests and three month-follow up. Plasma D-dimer (D-Di) is measured in case of low clinical probability. Helical computed tomography (CT) is performed in case of either high clinical probability or positive D-dimer. Lower limb venous compression ultrasonography (US) is done only in case of negative CT in a patient with a high clinical probability. Patients will be classified in two groups, as having or not having PE on predefined criteria according to the recent guidelines of the European Society of Cardiology by physicians who will be unaware of the SF assay result.

SF Assays. Soluble fibrin is measured by one site, using prototype assays, on both citrated and heparinized blood samples taken at baseline. Staff in charge of the assays are not aware of the clinical and diagnosis decisions.

Statistical Analysis of results. It will be performed independently by the Clinical Research Unit of Georges Pompidou European Hospital. The ROC curve will be built, the area under the curve will be calculated with its confidence interval. The most suitable threshold will be determined from the curve. Then the diagnostic performances of SF assay will be calculated according to the usual calculations.

Number of participants required. Taking into account an estimated area of 0.9 to 0.95 on preliminary data, the inclusion of 500 patients with suspected PE will allow calculation of the area under the ROC curve with an accuracy of 5%. This number will also allow calculation of the diagnostic performances of the SF assay with sufficient accuracy.

Duration of the study. The study period is three months for each patient, the total duration of the study is 28 months.

ELIGIBILITY:
Inclusion Criteria:

* patients are aged 18 years or older,
* outpatients from Emergency or Respiratory and Intensive Care Medicine Units,
* clinically suspected of PE

Exclusion Criteria:

* pregnant women,
* patients with contraindication to iodinated contrast media,
* patients treated with anticoagulants at curative doses,
* patients with suspected PE during hospitalization
* patients for which the three month-follow up is impossible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients from Emergency or Respiratory and Intensive Care Medicine Units, in a French Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Area under the ROC curve of the Soluble Fibrin for the diagnosis of PE | 28 months
  The ROC curve will be built, the area under the curve will be calculated with its confidence interval. The most suitable threshold will be determined from the curve.

SECONDARY OUTCOMES:
Threshold of the Soluble Fibrin assays for the diagnosis of PE | 28 months
  The most suitable threshold will be determined from the curve. Then the diagnosis performances of SF assays will be calculated according to the usual calculations.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Meyer, Ph D, Principal Investigator — Georges Pompidou European Hospital; Geneviève Contant, Ph D, Study Director — Diagnostica Stago R&D
Locations (1):
- Georges Pompidou European Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Roy PM, Colombet I, Durieux P, Chatellier G, Sors H, Meyer G. Systematic review and meta-analysis of strategies for the diagnosis of suspected pulmonary embolism. BMJ. 2005 Jul 30;331(7511):259. doi: 10.1136/bmj.331.7511.259. PMID 16052017
- [Background] Ginsberg JS, Siragusa S, Douketis J, Johnston M, Moffat K, Donovan D, McGinnis J, Brill-Edwards P, Panju A, Patel A, Weitz JI. Evaluation of a soluble fibrin assay in patients with suspected pulmonary embolism. Thromb Haemost. 1996 Apr;75(4):551-4. PMID 8743176
- [Background] Hetland O, Knudsen A, Dickstein K, Nilsen DW. Characteristics and prognostic impact of plasma fibrin monomer (soluble fibrin) in patients with coronary artery disease. Blood Coagul Fibrinolysis. 2002 Jun;13(4):301-8. doi: 10.1097/00001721-200206000-00005. PMID 12032395
- [Background] Mirshahi S, Soria C, Kouchakji B, Kierzek G, Borg JY, Varin R, Chidiac J, Drouet L, Mirshahi M, Soria J. New combinational assay using soluble fibrin and d-dimer determinations: a promising strategy for identifying patients with suspected venous thromboembolism. PLoS One. 2014 Mar 24;9(3):e92379. doi: 10.1371/journal.pone.0092379. eCollection 2014. PMID 24664182
- [Background] Konstantinides SV, Torbicki A, Agnelli G, Danchin N, Fitzmaurice D, Galie N, Gibbs JS, Huisman MV, Humbert M, Kucher N, Lang I, Lankeit M, Lekakis J, Maack C, Mayer E, Meneveau N, Perrier A, Pruszczyk P, Rasmussen LH, Schindler TH, Svitil P, Vonk Noordegraaf A, Zamorano JL, Zompatori M; Task Force for the Diagnosis and Management of Acute Pulmonary Embolism of the European Society of Cardiology (ESC). 2014 ESC guidelines on the diagnosis and management of acute pulmonary embolism. Eur Heart J. 2014 Nov 14;35(43):3033-69, 3069a-3069k. doi: 10.1093/eurheartj/ehu283. Epub 2014 Aug 29. No abstract available. PMID 25173341
- [Background] Klok FA, Mos IC, Nijkeuter M, Righini M, Perrier A, Le Gal G, Huisman MV. Simplification of the revised Geneva score for assessing clinical probability of pulmonary embolism. Arch Intern Med. 2008 Oct 27;168(19):2131-6. doi: 10.1001/archinte.168.19.2131. PMID 18955643
- [Background] Righini M, Van Es J, Den Exter PL, Roy PM, Verschuren F, Ghuysen A, Rutschmann OT, Sanchez O, Jaffrelot M, Trinh-Duc A, Le Gall C, Moustafa F, Principe A, Van Houten AA, Ten Wolde M, Douma RA, Hazelaar G, Erkens PM, Van Kralingen KW, Grootenboers MJ, Durian MF, Cheung YW, Meyer G, Bounameaux H, Huisman MV, Kamphuisen PW, Le Gal G. Age-adjusted D-dimer cutoff levels to rule out pulmonary embolism: the ADJUST-PE study. JAMA. 2014 Mar 19;311(11):1117-24. doi: 10.1001/jama.2014.2135. PMID 24643601